CLINICAL TRIAL: NCT03642002
Title: The Effects of Music Therapy on Adult Patients Requiring Mechanical Ventilation in the ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joanne Loewy, Director, Louis Armstrong Center for Music and Medicine at Mount Sinai Beth Israel, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 18-1079
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Hypoxemic Respiratory Failure; Acute Hypercapnic Respiratory Failure
Keywords: music therapy; song of kin; music medicine
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Intervention Model Description: Outcomes Assessor will be unfamiliar with desired outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Toning (Experimental): Vocal Tonal Holding
  Interventions: Other: Toning
- Ocean drum & SOK melody (Other): Ocean drum followed by melody of song of kin
  Interventions: Other: Ocean drum & SOK melody
- SOK (Experimental): Song of kin with lyric content
  Interventions: Other: SOK
- Process (Experimental): Processing of experience
  Interventions: Behavioral: Process
- Holding Harmonic Container (Experimental)
  Interventions: Other: Holding Harmonic Container

INTERVENTIONS:
Other: Toning — Music therapist will begin gentle breathing and toning on a descending "Ah" vowel to stimulate vibration in the chest and increase awareness of the breath. The patient will be encouraged to join the music therapist as is comfortable
  Arms: Toning
Other: Ocean drum & SOK melody — Music therapist will introduce ocean drum to mimic breathing sounds and will hum the melody of Song of Kin to begin entrainment process. Patient will be invited to join the music therapist in humming as is comfortable
  Arms: Ocean drum & SOK melody
Other: SOK — Music therapist will introduce sung lyric content of Song of Kin accompanied on guitar. Patient will be invited to sing with music therapist as is comfortable.
  Arms: SOK
Behavioral: Process — Music therapist will process patient experience and provide psycho-education on strategies for using music to promote comfort and enhance breath.
  Arms: Process
Other: Holding Harmonic Container — Music therapist will provide a holding harmonic container of IM7 - IVM7 and will improvise a repeating melody on "ah" based on the ambient sounds in the patient's immediate environment
  Arms: Holding Harmonic Container

SUMMARY:
While most studies in the medical literature that indicate "music" as an intervention may recognize its impact and capacity to decrease pain perception, anxiety, and/or its role in the regulation of cardiac and respiratory function in ICU patients, no identifiable studies have implemented entrained live music therapy protocols into clinical trials. Music therapy treatment is a non-pharmacological intervention that is individually tailored to the patient's needs and focuses on the assessment and intervention of a specific music application that is provided by a certified music therapist. Entrained music therapy focuses on a dynamic interaction between the patient and music therapist in which the music therapist attempts to promote relaxation and comfort through the patient's identified Song of Kin (SOK). This study measures the effects of live music therapy entrained to the vital signs of adult patients on duration of mechanical ventilation.

DETAILED DESCRIPTION:
The study will include 178 adult patients on mechanical ventilation. These patients will be randomly assigned to the music therapy group or control group and matched for diagnosis, co-morbidities, age, and gender. The music therapy group will utilize a certified music therapist to provide live music based on the patient's cultural preferences and entrainment. The primary outcome is a reduction in mechanical ventilation hours of 35% compared to the control group. Secondary outcomes include: Amount of sedation, Richmond Agitation-Sedation Scale (RASS), delirium and pain score, ICU and hospital length of stay. The researchers hypothesize that live entrained music therapy compared to control will result in a reduction in the time of extubation, amount of sedation administered, ICU and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acute hypoxemic respiratory failure, acute hypercapnic respiratory failure, and ARDS admitted to the ICU requiring mechanical ventilation
* Patients that are anticipated to remain on invasive mechanical ventilation for 48 hours or more will be screened for participation in the study

Exclusion Criteria:

* Under 18 years of age
* Identified hearing disorder
* Prior history of chronic respiratory failure requiring mechanical ventilation
* RASS score of -4, or -5
* Active seizures, or status epilepticus
* Cardiac arrest
* Coma
* End of life
* More than 2 vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative Length of Time on Ventilator | average 14 days

SECONDARY OUTCOMES:
Cumulative Length of Stay in Hospital | average 14 days
Respiration Rate | 15 minute intervals over 30 minute intervention
Heart Rate | 15 minute intervals over 30 minute intervention
Oxygen Saturation | 15 minute intervals over 30 minute intervention
Amount of sedation | 14 days
Richmond Agitation-Sedation Scale (RASS) | 14 days
  RASS is scored from +4 (combative) to -5 (unarousable), with lower score indicating more sedation.
State-Trait Anxiety Inventory (STAI) (Short Form) | 14 days
  To calculate the total STAI score (range 20-80):
  * Reverse scoring of the positive items (calm, relaxed, content) so 1=4, 2=3, 3=2, and 4=1;
  * Sum all six scores;
  * Multiply total score by 20/6
  * Scores are interpreted such that a "normal" score is approximately 24-36, Higher score indicates more anxiety
Confusion Assessment Method for the ICU (CAM-ICU) | 14 days
  CAM-ICU is a delirium monitoring instrument for ICU patients, scored for two possibilities: CAM-ICU Positive (where delirium is present for a patient) or CAM-ICU Negative (where delirium is not present for a patient).
Pain score | 14 days
  Numeric Pain Score (for enrollees able to speak). Pain score from 0 (no pain) to 10 (most pain)
Wong-Baker FACES ® Pain Rating Scale | 14 days
  Wong-Baker FACES ® Pain Rating Scale (for enrollees unable to speak). Pain score from 0 (no pain) to 10 (most pain)
ICU length of stay | average 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Loewy, DA, LCAT, MT-BC, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai West, New York, New York
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chlan LL. Psychophysiologic responses of mechanically ventilated patients to music: a pilot study. Am J Crit Care. 1995 May;4(3):233-8. PMID 7787918
- [Background] Canga B, Azoulay R, Raskin J, Loewy J. AIR: Advances in Respiration - Music therapy in the treatment of chronic pulmonary disease. Respir Med. 2015 Dec;109(12):1532-9. doi: 10.1016/j.rmed.2015.10.001. Epub 2015 Oct 19. PMID 26522499
- [Background] Chlan L. Effectiveness of a music therapy intervention on relaxation and anxiety for patients receiving ventilatory assistance. Heart Lung. 1998 May-Jun;27(3):169-76. doi: 10.1016/s0147-9563(98)90004-8. PMID 9622403
- [Background] Chlan LL. Music therapy as a nursing intervention for patients supported by mechanical ventilation. AACN Clin Issues. 2000 Feb;11(1):128-38. doi: 10.1097/00044067-200002000-00014. PMID 11040559
- [Background] Conti G, Mantz J, Longrois D, Tonner P. Sedation and weaning from mechanical ventilation: time for 'best practice' to catch up with new realities? Multidiscip Respir Med. 2014 Aug 29;9(1):45. doi: 10.1186/2049-6958-9-45. eCollection 2014. PMID 25473522
- [Background] Erdogan Z, Atik D. Complementary Health Approaches Used in the Intensive Care Unit. Holist Nurs Pract. 2017 Sep/Oct;31(5):325-342. doi: 10.1097/HNP.0000000000000227. PMID 28786890
- [Background] Hetland B, Lindquist R, Weinert CR, Peden-McAlpine C, Savik K, Chlan L. Predictive Associations of Music, Anxiety, and Sedative Exposure on Mechanical Ventilation Weaning Trials. Am J Crit Care. 2017 May;26(3):210-220. doi: 10.4037/ajcc2017468. PMID 28461543
- [Background] Hunter BC, Oliva R, Sahler OJ, Gaisser D, Salipante DM, Arezina CH. Music therapy as an adjunctive treatment in the management of stress for patients being weaned from mechanical ventilation. J Music Ther. 2010 Fall;47(3):198-219. doi: 10.1093/jmt/47.3.198. PMID 21275332
- [Background] Jaber S, Bahloul H, Guetin S, Chanques G, Sebbane M, Eledjam JJ. [Effects of music therapy in intensive care unit without sedation in weaning patients versus non-ventilated patients]. Ann Fr Anesth Reanim. 2007 Jan;26(1):30-8. doi: 10.1016/j.annfar.2006.09.002. Epub 2006 Nov 3. French. PMID 17085009
- [Background] Lee CH, Lee CY, Hsu MY, Lai CL, Sung YH, Lin CY, Lin LY. Effects of Music Intervention on State Anxiety and Physiological Indices in Patients Undergoing Mechanical Ventilation in the Intensive Care Unit. Biol Res Nurs. 2017 Mar;19(2):137-144. doi: 10.1177/1099800416669601. Epub 2016 Sep 21. PMID 27655993
- [Background] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Background] Loewy J, Hallan C, Friedman E, Martinez C. Sleep/sedation in children undergoing EEG testing: a comparison of chloral hydrate and music therapy. Am J Electroneurodiagnostic Technol. 2006 Dec;46(4):343-55. PMID 17285817
- [Background] Lindgren VA, Ames NJ. Caring for patients on mechanical ventilation: what research indicates is best practice. Am J Nurs. 2005 May;105(5):50-60; quiz 61. doi: 10.1097/00000446-200505000-00029. No abstract available. PMID 15867534
- [Background] Zilberberg MD, Shorr AF. Prolonged acute mechanical ventilation and hospital bed utilization in 2020 in the United States: implications for budgets, plant and personnel planning. BMC Health Serv Res. 2008 Nov 25;8:242. doi: 10.1186/1472-6963-8-242. PMID 19032766
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092